CLINICAL TRIAL: NCT04484142
Title: Phase 2, Single-arm, Open-label Study of DS-1062a in Advanced or Metastatic Non-small Cell Lung Cancer With Actionable Genomic Alterations and Progressed On or After Applicable Targeted Therapy and Platinum Based Chemotherapy (TROPION-Lung05)
Brief Title: Study of DS-1062a in Advanced or Metastatic Non-small Cell Lung Cancer With Actionable Genomic Alterations (TROPION-Lung05)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DS1062-A-U202; 2020-002774-27 (EudraCT Number)
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Metastatic Non-small Cell Lung Cancer; Advanced Metastatic Non-small Cell Lung Cancer; Non-small Cell Lung Cancer; DS-1062a; Datopotamab Deruxtecan
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DS-1062a 6.0 mg/kg (Experimental): Participants will receive 6.0 mg/kg of DS-1062a
  Interventions: Drug: DS-1062a

INTERVENTIONS:
Drug: DS-1062a — DS-1062a will be administered as an intravenous (IV) infusion once every 3 weeks
  Other Names: Datopotamab Deruxtecan

SUMMARY:
This is a study of the efficacy, pharmacokinetics, and safety of DS-1062a in participants with advanced or metastatic non-small cell lung cancer (NSCLC) with known actionable genomic alterations.

DETAILED DESCRIPTION:
This study will evaluate DS-1062a 6.0 mg/kg in participants with advanced or metastatic NSCLC with actionable genomic alterations and who have been previously been treated with 1 platinum-containing therapy and 1 or more lines of targeted therapy. The study will be divided into 3 periods: Screening Period, Treatment Period, and Follow-up Period. The primary analysis of Objective Response Rate (ORR) by blinded Independent Central Review (BICR) will be conducted after all participants either have been followed for at least 9 months after the start of study treatment or have discontinued from the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in the study must meet all inclusion criteria for this study.

* Sign and date the inform consent form (ICF) prior to the start of any study- specific qualification procedures.
* Adults ≥18 years (if the legal age of consent is >18 years old, then follow local regulatory requirements)
* Has pathologically documented NSCLC that:

  1. Has stage IIIB, IIIC, or stage IV NSCLC disease at the time of enrollment (based on the American Joint Committee on Cancer, Eighth Edition).
  2. Has one or more of the following documented activating genomic alterations: EGFR, ALK, ROS1, NTRK, BRAF, MET exon 14 skipping, or RET.

KRAS mutations in the absence of any of the genomic alterations specified above will be excluded.

Overexpression of EGFR, in the absence of activating mutations, is NOT sufficient for enrollment.

Participants who have not received osimertinib should be evaluated for the presence of EGFR T790M mutation after relapse/progression on/after the most recent EGFR tyrosine kinase inhibitor (TKI), unless the participant is already known to be positive with document results for this mutation or unless osimertinib is not locally approved.

* Has documentation of radiographic disease progression while on or after receiving the most recent treatment regimen for advanced or metastatic NSCLC.
* Participant must meet the following for advanced or metastatic NSCLC:

  1. Has been treated with at least one but no more than two cytotoxic agent-containing therapy in the metastatic setting:

     * One platinum-containing regimen (either as monotherapy or combination therapy).
     * May have received up to one additional line of cytotoxic agent-containing therapy.
     * Those who received a platinum-containing regimen as adjuvant therapy for early stage disease must have relapsed or progressed while on the treatment or within 6 months of the last dose OR received at least one additional course of platinum-containing therapy (which may or may not be same as in the adjuvant setting) for relapsed/progressive disease.
  2. May have received up to one checkpoint inhibitor (CPI)-containing regimen (may be in combination with a cytotoxic agent as part of a regimen described above or as an additional CPI regimen without a cytotoxic agent).
  3. Has been treated with 1 or more lines of non-CPI targeted therapy that is locally approved for the participant's applicable genomic alteration at the time of screening:

     * Those who received a targeted agent for the applicable genomic alterations in the study as adjuvant therapy for early stage disease must have relapsed or progressed while on the treatment or within 6 months of the last dose OR received at least one additional course of targeted therapy for the same genomic alterations (which may or may not be same agent used in the adjuvant setting) for relapsed/progressive disease.
     * Participants who have been treated with a prior TKI must receive additional targeted therapy, if clinically appropriate, for the genomic alterations that are considered amenable or the participant will not be allowed in the study.
* Must undergo a mandatory pre-treatment tumor biopsy procedure or if available, a tumor biopsy that was recently collected (within 3 months of screening) after completion of the most recent anticancer treatment regimen and that has a minimum of 10 × 4 micron sections or a tissue block equivalent of 10 × 4 micron sections may be substituted for the mandatory biopsy collected during screening.
* Measurable disease based on local imaging assessment using RECIST v1.1.
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 - 1 at screening.

Exclusion Criteria:

Participants meeting any exclusion criteria for this study will be excluded from this study.

* Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with clinically inactive brain metastases may be included in the study.
* Has leptomeningeal carcinomatosis.
* Has prior treatment with:

  1. Any chemotherapeutic agent targeting topoisomerase I, including antibody drug conjugate (ADC) containing such agent.
  2. TROP2-targeted therapy.
* Uncontrolled or significant cardiovascular disease:

  1. History of myocardial infarction within 6 months prior to Cycle 1 Day 1.
  2. History of uncontrolled angina pectoris within 6 months prior to Cycle 1 Day 1.
  3. Symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV) at screening. Participants with a history of Class II to IV CHF prior to screening must have returned to Class I CHF and have LVEF ≥50% (by either an ECHO or MUGA scan within 28 days of Cycle 1 Day 1) in order to be eligible.
  4. History of serious cardiac arrhythmia requiring treatment.
  5. LVEF <50% or institutional lower limit of normal by ECHO or MUGA scan.
  6. Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg).
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Clinically significant corneal disease.
* Has other primary malignancies, except adequately resected non-melanoma skin cancer, curatively treated in situ disease, or other solid tumors curatively treated, with no evidence of disease for ≥3 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2025-12-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (84):
- United States (28):
  - Mayo Clinic, Phoenix, Arizona
  - University of California San Diego, La Jolla, California
  - UCLA, Santa Monica, California
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Sarah Cannon Research Institute at Florida Cancer Center, North, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Sarah Cannon Research Institute at Florida Cancer Center, South, Port Charlotte, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - The Office of Dr. Frederick P. Smith MD, Chevy Chase, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - XCancer / Regional Cancer Care Associate (Astera), East Brunswick, New Jersey
  - NYU Langone Medical Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - New York Cancer and Blood Specialists, Port Jefferson, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Avera Cancer Institute Sioux Falls, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute at Tennessee Oncology - Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Athens, Virginia
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
- France (9):
  - APHM - Hopital Nord, Marseille, Bouches-Du-RhÃ´ne
  - University Hospital of Nantes, Nantes, Loire-Atlantique
  - CHU Toulouse Hopital Larrey, Toulouse, Occitanie
  - Centre Leon Berard, Lyon, Rhone
  - CHU Louis Pradel, Lyon
  - Institut Curie, Paris
  - Hopitaux Universitaire de Strasbourg- Nouvel Hopital Civil, Strasbourg
  - Centre Hospitalier Intercommunal Toulon La Seyne sur mer Hopital Sainte-Musse, Toulon
  - Gustav Roussy Cancer Campus Grand Paris, Villejuif, Île-de-France Region
- Germany (6):
  - Thoraxklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Asklepios Fachklinik Muenchen-Gauting, Gauting, Bavaria
  - IKF Krankenhaus Nordwest, Frankfurt am Main, Hesse
  - Universitaet zu Koeln - Uniklinik Koeln, Cologne, North Rhine-Westphal
  - Medizinische Hochschule Hannover, Hanover
  - Thoraxklinik Heidelberg gGmbH, Heidelberg
- Hungary (2):
  - National Koranyi Institute for TB and Pulmonology, Budapest
  - Pulmonology Hospital Törökbálint, Törökbálint
- Italy (8):
  - Azienda Ospedaliera Universitaria Policlinico-OVE, Catania, CT
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, RM
  - University of Turin San Luigi Hospital, Orbassano, Torino
  - Azienda Ospedaliero-Universitaria S. Orsola Malpighi, Bologna
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliera Arcispedale Santa Maria, Reggio Emilia
- Japan (14):
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kyoto University Hospital, Kyoto, Kyoto
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka City General Hospital, Osaka, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - Kindai University Hospital, Ōsaka-sayama, Osaka
  - Shizuoka Cancer Center, Nagaizumi-chō, Shizuoka
  - Tokushima University Hospital, Tokushima, Tokushima
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo
  - Aichi Cancer Center Hospital, Aichi
- Netherlands (2):
  - The Netherlands Cancer Institute, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
- South Korea (5):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda, Madrid
  - Hospital Regional Universitario Malaga, Málaga, Malaga
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario Vall dHebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital NTUH, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: http://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Sands J, Ahn MJ, Lisberg A, Cho BC, Blumenschein G Jr, Shum E, Pons Tostivint E, Goto Y, Yoh K, Heist R, Shimizu J, Lee JS, Baas P, Planchard D, Perol M, Felip E, Su WC, Zebger-Gong H, Lan L, Liu C, Howarth P, Chiaverelli R, Paz-Ares L. Datopotamab Deruxtecan in Advanced or Metastatic Non-Small Cell Lung Cancer With Actionable Genomic Alterations: Results From the Phase II TROPION-Lung05 Study. J Clin Oncol. 2025 Apr;43(10):1254-1265. doi: 10.1200/JCO-24-01349. Epub 2025 Jan 6. PMID 39761483

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 137 participants who met all inclusion criteria and no exclusion criteria were enrolled to receive Dato-DXd treatment in 50 clinical sites, North America= 15, Europe= 14, Asia Pacific= 21.
Groups:
- Dato DXd 6.0 mg/kg Q3W: Participants received an intravenous (IV) infusion of Dato DXd administered at a dose of 6.0 mg/kg every 3 weeks (Q3W) on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | Dato DXd 6.0 mg/kg Q3W
Started | 137
Completed | 20
Not Completed | 117
Not completed — Adverse Event | 13
Not completed — Progressive Disease | 87
Not completed — Clinical Progression | 10
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The baseline demographic characteristics were assessed in the Full Analysis Set, which includes all subjects who received at least 1 dose of study drug.
Arm/Group | Dato DXd 6.0 mg/kg Q3W
Number analyzed (Participants) | 137
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 91
  >=65 years | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (11.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83
  Male | 54
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 78
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 43
  More than one race | 15
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response Rate (ORR) Based on Blinded Independent Central Review (BICR)
Description: ORR is defined as the proportion of participants with a best overall response of confirmed complete response (CR) or confirmed partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Time Frame: From baseline until disease progression, death, or other protocol defined reason, up to approximately 24 months.
Population: Outcome Measure was assessed in the Full Analysis Set, which includes all subjects who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dato DXd 6.0 mg/kg Q3W
Number analyzed (Participants) | 137
percentage of participants | 35.8 [27.8 to 44.4]

2. Secondary Outcome: Duration of Response (DOR)
Time Frame: From baseline up to approximately 24 months
Reporting Status: Not Posted, anticipated posting 2027-05

3. Secondary Outcome: Progression-free Survival (PFS)
Time Frame: From baseline up to approximately 24 months
Reporting Status: Not Posted, anticipated posting 2027-05

4. Secondary Outcome: Overall Survival (OS)
Time Frame: From baseline up to approximately 24 months
Reporting Status: Not Posted, anticipated posting 2027-05

5. Secondary Outcome: Pharmacokinetic Parameter Maximum Concentration (Cmax)
Time Frame: From baseline up to approximately 24 months
Reporting Status: Not Posted, anticipated posting 2027-05

6. Secondary Outcome: Pharmacokinetic Parameter Time to Maximum Concentration (Tmax)
Time Frame: From baseline up to approximately 24 months
Reporting Status: Not Posted, anticipated posting 2027-05

7. Secondary Outcome: Pharmacokinetic Parameter Area Under the Concentration-Time Curve (AUC)
Time Frame: From baseline up to approximately 24 months
Reporting Status: Not Posted, anticipated posting 2027-05

8. Secondary Outcome: Percentage of Participants Who Reported Treatment-emergent Adverse Events (TEAE)
Time Frame: From baseline up to approximately 24 months
Reporting Status: Not Posted, anticipated posting 2027-05

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected from the date of first treatment, up to 24 months.
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event with a start or worsening date on or after the start of study treatment until 35 days since the last dose of study treatment.
Arm/Group | Dato DXd 6.0 mg/kg Q3W
All-Cause Mortality (participants affected / at risk) | 68/137
Serious Adverse Events (participants affected / at risk) | 34/137
Other Adverse Events (participants affected / at risk) | 135/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dato DXd 6.0 mg/kg Q3W (N=137)
Cataract (Eye disorders) | 1 (2)
Glaucoma (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastric perforation (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Fatigue (General disorders) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dato DXd 6.0 mg/kg Q3W (N=137)
Anaemia (Blood and lymphatic system disorders) | 21 (24)
Dry eye (Eye disorders) | 15 (16)
Vision blurred (Eye disorders) | 12 (12)
Keratitis (Eye disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 82 (117)
Stomatitis (Gastrointestinal disorders) | 79 (89)
Constipation (Gastrointestinal disorders) | 43 (47)
Vomiting (Gastrointestinal disorders) | 31 (41)
Diarrhoea (Gastrointestinal disorders) | 17 (19)
Fatigue (General disorders) | 34 (40)
Asthenia (General disorders) | 21 (35)
Pyrexia (General disorders) | 14 (17)
Malaise (General disorders) | 11 (13)
Oedema peripheral (General disorders) | 7 (7)
COVID-19 (Infections and infestations) | 20 (20)
Infusion related reaction (Injury, poisoning and procedural complications) | 9 (9)
Weight decreased (Investigations) | 14 (14)
Amylase increased (Investigations) | 12 (17)
Aspartate aminotransferase increased (Investigations) | 9 (9)
Blood creatinine increased (Investigations) | 9 (12)
White blood cell count decreased (Investigations) | 9 (13)
Alanine aminotransferase increased (Investigations) | 8 (10)
Neutrophil count decreased (Investigations) | 8 (10)
Blood alkaline phosphatase increased (Blood and lymphatic system disorders) | 7 (8)
Decreased appetite (Metabolism and nutrition disorders) | 37 (44)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (10)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Headache (Nervous system disorders) | 14 (14)
Dizziness (Nervous system disorders) | 9 (9)
Dysgeusia (Nervous system disorders) | 8 (8)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (16)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 70 (71)
Rash (Skin and subcutaneous tissue disorders) | 21 (27)
Pruritus (Skin and subcutaneous tissue disorders) | 14 (14)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT04484142/Prot_SAP_000.pdf